CLINICAL TRIAL: NCT02932098
Title: Post-Op Gynecological Oncology Web-Based App Study
Brief Title: Post-Operative Gynecological Oncology App Study
Acronym: POGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: University of Tennessee West Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-04470XP R073237324
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Genital Neoplasm, Female
MeSH Terms: conditions — Genital Neoplasms, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- App Notifications (Experimental): The web-based app will be used to remind patients of discharge instructions, ask questions related to current prescription pain medication use, new symptoms, or changes in the severity of symptoms. Patients will receive reminders via text or email to use the app. Daily reminders will be sent in Week 1, every other day in Week 2, and once per week for Weeks 3-4. All participants will be followed for a minimum of 30 days and will be asked to complete a baseline survey at enrollment and a follow-up survey scheduled 30 days after hospital discharge.
  Interventions: Behavioral: Discharge instructions reminders; Behavioral: Prompts to report symptoms via the web-enabled app; Behavioral: Clinical Alerts
- Usual Care (Active Comparator): Patients will have access to the web-based app, but will not receive reminders to use it. All participants will be followed for a minimum of 30 days and will be asked to complete a baseline survey at enrollment and a follow-up survey scheduled 30 days after hospital discharge.
  Interventions: Behavioral: Clinical Alerts

INTERVENTIONS:
Behavioral: Discharge instructions reminders — Week 1, Day 1: Click through each discharge instruction; Week 1, Days 2-7: Click through single list of all discharge instructions.
  Participants will receive a reminder of discharge instructions everyday for the first week post-discharge.
  Arms: App Notifications
Behavioral: Prompts to report symptoms via the web-enabled app — Group will receive reminders to enter new symptoms or changes in symptoms (based on a Likert scale or Y/N) on the following schedule: Week 1 (daily), Week 2 (every other day), Weeks 3-4 (once per week)
  Arms: App Notifications
Behavioral: Clinical Alerts — Alerts based on certain response thresholds are generated to inform the patient's care team of any concerning responses or trends that emerge from the patient reported outcomes. These alerts will inform providers of particular patient-related adverse events or symptoms requiring an intervention prior to the point that emergent medical care is needed. Information in the alert emails will include the participant's Medical Reference Number (MRN), initials, date of birth, and details about the symptom(s) that generated the alert. Pod nurses instructed to respond to any clinical alerts (sent via email) as soon as possible following standard of care.

SUMMARY:
Purpose: The purpose of this study will be to test the use of a web-based mobile application (app) initiated at the time of hospital discharge to engage and monitor patients in order to efficiently deliver better outcomes. The mobile app will be used to remind patients of discharge instructions, assess adherence treatment regimens, and evaluate symptoms.

Rationale: Approximately 60% of patients with ovarian cancer have advanced stage disease at diagnosis, and thus aggressive surgical procedures are often medically necessary. Recent evidence suggests that nearly one in five patients hospitalized for ovarian cancer surgery will be readmitted within 30 days of discharge. Patients readmitted within 30 days have a 50% increase in one-year mortality rates and significantly increased costs of care. In addition, many of the conditions and complications that led to readmission could potentially have been avoided with more intensive post-surgical follow-up care. Mobile health technologies can effectively and efficiently connect patients with their healthcare team and have been shown to improve treatment adherence and reduce avoidable ER visits and hospitalizations.

DETAILED DESCRIPTION:
The investigators plan to enroll 15 subjects per study arm, for a total of 30 participants. Potential subjects for recruitment will be identified from the electronic health records system of the West Cancer Center. The West Cancer Center employs four physicians specializing in gynecologic oncology who account for nearly 100% of open abdominal hysterectomies among ovarian cancer patients in the region. All four physicians have expressed strong support of the study and have agreed to actively participate by allowing screening of electronic health record data to identify appropriate patients and referral of eligible patients to the Nurse Coordinator for possible consent. The Nurse Coordinator will approach eligible patients during their surgery planning visit or in the hospital prior to surgery to provide an overview of the research study and seek informed consent.

Patients who provide informed consent will immediately be asked to complete a brief baseline survey about their preferences for receiving prompts, either via email or via cell phone using a text message. After survey administration, all patients will be registered in the mobile health app, which will be used provide discharge care instructions and monitor their progress upon discharge. Study participants will then be randomized into one of two arms: 1) active prompts to use the study app or 2) use of study app, but no prompts. All participants will be followed for a minimum of 30 days and will be asked to complete a follow-up survey during a scheduled in-clinic appointment at the end of the study.

Baseline and follow-up questionnaires will collect data on quality of life (SF-12), physical symptoms, activities of daily life, prescription narcotic use, health literacy, demographics and use of health care services (e.g. ER visit, hospital admission, clinic appointment). The web-based app will be used to remind patients of discharge instructions, ask questions related to current prescription pain medication use, new symptoms, or changes in the severity of symptoms.

Data from this study will be derived from the following sources: electronic health data to capture treatment changes and disease severity; responses to baseline and follow-up questionnaires to measure self-reported behaviors, including quality of life, use of prescription pain medication and care utilization; and post-study semi-structured interviews with physicians and patients to provide qualitative feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (age≥18)
2. Diagnosed (or suspected) of ovarian, fallopian, or primary peritoneal cancer (any stage)
3. Scheduled for open abdominal surgery for cancer diagnosis and/or staging during recruitment period
4. Have a mobile device with a data plan or a home computer with Internet
5. Have a valid email address
6. Willing to complete brief symptom reports on the app in the 30 days following hospital discharge

Exclusion Criteria:

1. Unable to communicate in English
2. A concomitant diagnosis of endometrial or breast cancer
3. Did not have open abdominal surgery for a hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Improve quality of life (SF-12) | 30 days
  The primary data analysis will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure changes in quality of life from baseline and at 30-days, and compare changes between the two study arms.

SECONDARY OUTCOMES:
Reduce re-admission and emergency department visits to the hospital within 30-days of discharge | 30 days
  Investigators also plan to carry out a secondary analysis, which will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure any healthcare utilization within the 30 day post-discharge, and compare utilization between the two study arms.
Activities of daily living, status 30 days after discharge | 30 days
  Investigators also plan to carry out a secondary analysis, which will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure participants' independence 30 days post-discharge using an Activities of Daily Living (ADL) assessment adapted from the Katz Index of Independence, and compare status between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Graetz, PhD, Principal Investigator — University of Tennessee
Locations (3):
- United States (3):
  - West Cancer Center, DESOTO, 7668 Airways Blvd., Southaven, Mississippi
  - West Cancer Center, MIDTOWN, 1588 Union Ave., Memphis, Tennessee
  - West Cancer Center, EAST MEMPHIS, 7945 Wolf River Blvd, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided